CLINICAL TRIAL: NCT00012909
Title: Development and Evaluation of a Hormone Replacement Therapy Decision-Aid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: PCC 98-039
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-11

CONDITIONS: Menopause; Hormone Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Behavioral: Hormone Replacement Therapy Decision-Aid

INTERVENTIONS:
Behavioral: Hormone Replacement Therapy Decision-Aid

SUMMARY:
The decision regarding the use of post-menopausal estrogen hormone replacement therapy (HT) is complex because patients must balance the short and long-term risks and benefits. Information from new and important clinical trials must also be considered. The purpose of this research is to develop and evaluate the efficacy of a HT CD-ROM decision-aid in improving the decision making process for women considering the use of estrogen HT.

DETAILED DESCRIPTION:
Background:

The decision regarding the use of post-menopausal estrogen hormone replacement therapy (HT) is complex because patients must balance the short and long-term risks and benefits. Information from new and important clinical trials must also be considered. The purpose of this research is to develop and evaluate the efficacy of a HT CD-ROM decision-aid in improving the decision making process for women considering the use of estrogen HT.

Objectives:

The objectives of the study are to: 1) develop a model of the decision-making process for postmenopausal women considering hormone (HT), based on Multi-Attribute Utility Theory (MAUT); 2) produce an interactive CD-ROM decision-aid for HT; 3) evaluate the effect of the interactive CD-ROM decision-aid on patient satisfaction with decision (SWD) and knowledge about menopause and HT; and 4) test the effect of the interactive CD-ROM decision-aid on women�s decisions regarding use of HT.

Methods:

Phase I (completed) used structured interviews and surveys in the development of a decision model for HT. In phase II, an interactive CD-ROM decision-aid was developed and a randomized controlled trial (RCT) of its effect on decision processes was conducted. Postmenopausal women, aged 45-74 were recruited from the primary care clinics of the four participating Veterans Affairs hospitals: Milwaukee, Madison, Chicago-Hines, and Chicago-Westside. The primary hypothesis was that women who use the CD-ROM decision-aid would demonstrate increased satisfaction with their decision regarding hormone replacement therapy use compared to women receiving the control intervention.

Status:

Enrollment and follow-up assessments have been completed. The study is in the analysis phase. The study was presented to the VA HSR&D Combined Monitoring Board on February 5, 2003 and the committee voted unanimously to recommend continuation of the trial. The study has had one publication and several scientific abstract presentations.

ELIGIBILITY:
Inclusion Criteria:

- postmenopausal as defined by: Amenorrhea for 12 months or FSH greater than or equal to 25

Exclusion Criteria:

* unable to speak English
* are assessed not to have capacity for making medical decisions for their own care
* had alcohol or drug abuse issues in past 6 months before baseline visit
* personal history of breast cancer, active liver disease, active vascular thrombosis, and/or active unexplained vaginal bleeding

Ages: 45 Years to 74 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Study Completion 2004-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn M. Schapira, MD MPH, Principal Investigator — Clement J. Zablocki VA Medical Center, Milwaukee, WI; Arneda Van White, MD, Principal Investigator — Edward Hines Jr. VA Hospital, Hines, IL
Locations (3):
- United States (3):
  - Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois
  - Clement J. Zablocki VA Medical Center, Milwaukee, WI, Milwaukee, Pennsylvania
  - William S. Middleton Memorial Veterans Hospital, Madison, WI, Madison, Wisconsin

REFERENCES:
- [Result] Schapira MM, Gilligan MA, McAuliffe TL, Nattinger AB. Menopausal hormone therapy decisions: insights from a multi-attribute model. Patient Educ Couns. 2004 Jan;52(1):89-95. doi: 10.1016/s0738-3991(02)00266-5. PMID 14729295